CLINICAL TRIAL: NCT05729841
Title: StORMM 1:What Effect Does Rowing 3000 Miles Across Atlantic Ocean Have on Calf Muscle Size? StORMM 2. In the Catabolic State of Extreme Endurance, is Muscle Loss Uniform or Can the Human Body Select Depending on Load and Nutrient Availability?
Brief Title: Study of Ocean Rowing Muscle Metabolism. 1. What Effect Does Rowing 3000 Miles Across Atlantic Ocean Have on Calf Muscle Size? 2. In the Catabolic State of Extreme Endurance, is Muscle Loss Uniform or Can the Human Body Select Depending on Load and Nutrient Availability?
Acronym: StORMM
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 201021-A-08
Record Dates: First submitted 2023-01-16; First posted 2023-02-15 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Exercise
Keywords: ocean rowing; ultra endurance; doubly labelled water
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ocean row — the Talisker Whisky Atlantic Challenge annual ocean rowing race.

SUMMARY:
Little is known on the human adaptation to extreme endurance and with the increasing popularity in long duration events we seek to provide insight into the physiological and metabolic adaptation processes of ocean rowing.

Rowing 12-18 hours a day will illicit a high energy expenditure and anecdotally people have lost large amounts of body weight and variable amounts of muscle mass, particularly in the lower limbs. This may provide insights and a potential new model to to study muscle unloading.

DETAILED DESCRIPTION:
Previous research has investigated factors determining muscle loss through bed rest and limb immobilisation. These methods are limited in that some do not include inflammation or changes in nutrition, which have been shown to be key drivers of muscle loss. These studies aim to investigate a potentially new model of muscle unloading.

Ocean rowing is an ultra-endurance sport where people spend 35-90 days at sea. Usually rowing for a minimum of 12 hours a day, in a 2-hour on/off shift pattern with daily food rations. Rowers lose body and muscle mass. There is likely to be low-grade inflammation, nutritional deficit, fatigue and rowers do not stand up for the entire crossing. Part 1 aims to quantify this muscle loss by inviting rowers in the annual 3000 mile Talisker Whisky Atlantic Challenge 2020 to take part. While part 2 aims to continue the work by measuring upper and core muscles as well as lower limb muscles from the first study with the aim of understanding how the body allocates resources in a hypocaloric, high energy expenditure environment.

Muscle mass of the lower limbs of the rowers will be measured with ultrasound, as well as body mass, body composition, energy expenditure and nutritional intake, the week before the race and immediately after arrival in Antigua. As well as adding novel insights to the knowledge base around factors affecting ultra endurance performance, the results will then be used to inform future intervention studies aimed at preventing muscle loss.

ELIGIBILITY:
Inclusion Criteria:

- Taking part in the Talisker Whisky Atlantic Challenge 2020 and 2021

Exclusion Criteria:

- lower limb amputee musculoskeletal, metabolic, neurological disease pacemaker fitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, fit and active males and females aged 18 and over
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | 5-7 days in final week of row
  Amount of kcals expended per day
Calf Muscle thickness | 5-7 weeks
  Pre - Post measurements of calf muscle thickness
Energy Intake | 5-7 days in final week of row
  Amount of kcals consumed per day

SECONDARY OUTCOMES:
Difference in rate of muscle thickness loss between males and females | 5-7 weeks
  Absolute and relative differences in energy balance, body mass loss or muscle loss
Difference in rate of muscle thickness loss in older vs younger rowers | 5-7 weeks
  Are there any age-related differences in energy balance, body mass loss or muscle loss

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD